CLINICAL TRIAL: NCT06620588
Title: Perioperative Outcomes of a Prehabilitation Programme for Surgical Patients Undergoing Major Surgery: a Pilot Interventional
Brief Title: PREPARE-M 2024 Undergoing Major Surgery: a Pilot Interventional
Status: Recruiting | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PREPARE24
Record Dates: First submitted 2024-08-11; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Prehabilitation
Keywords: Prehabilitation; frail; elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PREPARE: Patients will receive the routine preoperative physiotherapy assessment, nutrition education, exercise instructions, and inspiratory muscle training if their maximal inspiratory pressure (MIP) is less than100 cmH2O. These sessions, lasting 20 to 40 minutes, will include physiotherapy education and instructions for a home-based, unsupervised exercise program.
  Additionally, patients will undergo study-related measurements of baseline MIP using a handheld digital manometer, the 6-minute walk test (6MWT), handgrip strength (HGS) of the dominant hand, and 30-second and 1-minute Sit-To-Stand (STS) tests.

SUMMARY:
Study plan to conduct a pilot interventional study to evaluate the impact of a prehabilitation program on physical function and clinical outcomes. The prehabilitation program will include preoperative physiotherapy assessment, nutrition education, exercise instructions, and inspiratory muscle training for patients with MIP<100 cmH2O. Currently, Singapore General Hospital offers the "Prehabilitation for Elderly Frail Patients Undergoing Elective Surgeries (PREPARE)" program, targeting frail patients undergoing major surgery. The primary outcome of the study is the change in physical function, measured by handgrip strength (HGS), from baseline to 3 days before surgery. Secondary outcomes include changes in the 6-minute walk test (6MWT), maximal inspiratory pressure (MIP), and sit-to-stand (STS) parameters from baseline to 3 days before surgery and 4-5 weeks postoperatively. Additionally, study will also assess postoperative complications (using the Comprehensive Complication Index), postoperative morbidity (using the Postoperative Morbidity Survey), length of hospital stay (LOS), and Health-Related Quality of Life (HRQoL) outcomes.

DETAILED DESCRIPTION:
The exercise instructions given in the PREPARE program are part of the standard treatment and care is taken to ensure that the exercises are done safely at home. The only research segment is measurement of the parameters and clinical outcomes."

Patient Visits: 1. Recruitment/Enrollment (Visit 1 - coincide with PAC visit) Once informed consent is obtained. Patients will have the following measurements taken.

1. Baseline Maximal Inspiratory Pressure (MIP) using a handheld digital manometer,
2. 6-minute walk test (6MWT),
3. handgrip strength (HGS) of the dominant hand, and
4. 30s and 1-minute Sit-To-Stand (STS).

In addition, all patients will receive the routine (20 - 40 minutes) preoperative physiotherapy education, home exercise instructions and inspiratory muscle training (if MIP < 100 cmH2O).

2. Follow up (Phone call) Patients will receive follow-up phone calls once weekly to check if they have any problems following the home exercise instructions given to them on visit 1.

3. Follow up (Visit 2) - Pre-Op (3 days before Operation) Patients will have the measurements taken again.

4. Follow up (Visit 3) - Between 4 to 5 weeks post-operation. Patients will have the measurements taken again.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 65 years who are undergoing elective major non-cardiac surgery
* Edmonton Frail Score (EFS) of 6 or higher

Exclusion Criteria:

* Patients who are unable to provide written informed consent

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elective surgery patients , coming in for their pre-admission assessments
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The change in physical function between baseline and 3 days prior to surgery as measured by the handgrip strength | Baseline
  The change in physical function between baseline and 3 days prior to surgery as measured by the handgrip strength (HGS). HGS is a recognized marker of overall muscle and physical function and was chosen because it can be easily obtained from most frail elderly patients in our non-cardiac surgical population and is not limited by factors such as lower limb weakness, pain, or lower limb amputations.

SECONDARY OUTCOMES:
Change in 6-minute walk test (6MWT) from baseline to day of surgery to postoperatively 6MWT | Baseline, 3 days prior to surgery and between 4-5 weeks postoperatively
  6MWT correlates moderately with anaerobic threshold and low preoperative 6MWT values have been associated with increased odds of developing postoperative pulmonary complications and poorer health-related quality of life in physical domains.
Change in functional parameters : handgrip strength | baseline, 3 days prior to surgery and between 4-5 weeks postoperatively
30-day postoperative complications that will be assessed using the Comprehensive ComplicationIndex (CCI) | Up to 30 days after operation
Change in Health Related Quality of Life (HRQoL) outcomes, measured by the EQ-5D-3L, pre and post-operatively. | Baseline and pre-operation (4-5 weeks after op)
  0-100 , 0 as the worse imaginable health state to the best imaginable health state
30-day postoperative complications that will be assessed using the Postoperative Morbidity Survey (POMS) | Up to 30 days after operation
Change in functional parameters 30s and 1-min Sit to stand | baseline, 3 days prior to surgery and between 4-5 weeks postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore